CLINICAL TRIAL: NCT06278194
Title: Change of the Masseter Muscle Thickness Measured by Ultrasonography After Gasser Ganglion Radiofrequency Thermocoagulation Treatment
Brief Title: Masseter Muscle Thickness in Gasser Ganglion Radiofrequency Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Erken, Medical doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.11.2023.589
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Trigeminal Neuralgia; Gasserian Ganglion; Lesion
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated with gasserian ganglion RFT for trigeminal neuralgia (Other): In patients who have undergone radiofrequency thermocoagulation (RFT) of the gasserian ganglion for the treatment of trigeminal neuralgia, the thickness of the masseter muscle will be measured bilaterally, free and contracted, by ultrasound on the day of the procedure (just before the procedure) and at 1 and 3 months after the procedure.
  Interventions: Procedure: Gasserian Ganglion Radiofrequency Thermocoagulation

INTERVENTIONS:
Procedure: Gasserian Ganglion Radiofrequency Thermocoagulation — Gasserian ganglion radiofrequency thermocoagulation is performed in the operating room under fluoroscopy. In sterile condition, the foramen ovale is shown by the pain management specialist under fluoroscopy guidance. After this condition, the entry of the needle is marked and anaesthetised with local anaesthetic. After the entry of the gasserian ganglion with the radiofrequency needle, 10 cm long, the location is checked with sensory and motor stimulation. If the placement is correct, 70 degrees 70 seconds of radiofrequency thermocoagulation is applied.

SUMMARY:
Trigeminal neuralgia is common painful disorder in pain medicine clinics. Gasserian ganglion radiofrequency thermocoagulation is one of the treatment option in patients with trigeminal neuralgia in refractory cases. The most commonly involved branch in trigeminal neuralgia is the mandibular branch. Masseter muscle is innervated by mandibulary nerve branch of the trigeminal nerve.

The radiofrequency thermocoagulation therapy is used to ablate the affected trigeminal nerve branch and some of patients complain of subjective masseter weakness after this procedure.

In theoretical basis, muscles innervated by target nerve are affected from ablation procedure. In this study the primary aim is to evaluate the change of the masseter muscle thickness in patients treated by gasserian ganglion radiofrequency thermocoagulation. The results may also show possible functional effect of the procedure related with masseter muscle.

ELIGIBILITY:
Inclusion Criteria:

* Pain refractory to medical therapy for at least 3 months
* Planning radiofrequency thermocoagulation of gasserian ganglion
* Accept ultrasound measurements to be performed

Exclusion Criteria:

* Refused to participate in the study
* Not attending follow-ups regularly
* Coagulation disorder
* Pregnancy
* Localized or systemic infection

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Masseter muscle thickness | Pre-procedural time
  The thickness of the masseter muscle will be measured and recorded by ultrasound while bilaterally contracted and relaxed.
Masseter muscle thickness | Post-procedural first month
  The thickness of the masseter muscle will be measured and recorded by ultrasound while bilaterally contracted and relaxed.
Masseter muscle thickness | Post-procedural third month
  The thickness of the masseter muscle will be measured and recorded by ultrasound while bilaterally contracted and relaxed.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Tanyel Saraçoğlu, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)